CLINICAL TRIAL: NCT02881047
Title: Ablative Fractional Laser Resurfacing for the Treatment of Scars and Contractures Caused by Sclerotic Skin Changes Chronic Graft Versus Host Disease
Brief Title: Ablative Fractional Laser for Sclerotic GVHD-Associated Joint Contractures
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: UPCC 14613
Record Dates: First submitted 2016-08-24; First posted 2016-08-26 (Estimated); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Subjects With Severe, Refractory Sclerotic Skin Changes
MeSH Terms: interventions — Lasers, Gas; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rAblative Fractional Laser for Sclerotic GVHD-Associated Joint (Experimental): Range of motion limitations and joint contractures due to sclerotic GVHD across a specific joint / limb"
  Interventions: Device: CO2 Laser; Radiation: Ultrasound; Diagnostic Test: Skin Biopsy

INTERVENTIONS:
Device: CO2 Laser — Perform ablative fractional resurfacing using a 10,600nm carbon dioxide (CO2) laser targeted to thickened, sclerotic plaques causing range of motion limitation and contracture across joints.
Radiation: Ultrasound — Patients will undergo ultrasound of the planned treatment site to measure skin thickness and blood flow via Doppler ultrasound.
Diagnostic Test: Skin Biopsy — standard 4mm punch biopsy of the skin at the planned treatment site for histologic assessment of skin thickness and sclerosis.

SUMMARY:
Graft versus host disease (GVHD) is a common complication of allogeneic stem cell transplant.Chronic GVHD is characterized by skin thickening and tightening. Advanced sclerosis can lead to reduced range of motion and incapacitating joint contractures. Once present, there are few therapeutic options. We will treat sclerosis and limb contractures with an ablative fractional laser, a device FDA-approved for scar treatment. This approach has successfully treated contracturesdue to burn scars.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able to give informed consent
* All adult patients (18 years of age or older) Severe sclerotic skin changes of chronic graft versus host disease meeting a score of 3 on the NIH consensus criteria for organ scoring of chronic GVHD,
* a score defined by deep sclerotic features with hidebound skin which cannot be pinched together, resulting in impaired motion.
* According to the NIH criteria, the patient need not have widespread cutaneous GVHD; hidebound skin OR impaired mobility receive a score of 3 (highest score).
* Demonstrable range of motion limitations and joint contractures due to sclerotic GVHD across a specific joint / limb amenable to laser therapy must be present. - - Patients must note an inability to bend the joint (e.g. foot, wrist, elbow) freely which compromises the ability to perform specific tasks (e.g. walking up or down stairs, grabbing / making a fist, lifting or raising thearms over the head). As these functional limitations are by their nature subjective (and NIH scoring criteria are themselves subjective) determination of eligibility will be made by the investigator.
* ECOG Performance Status shall be 0-3

Exclusion Criteria:

* Persons unable to provide informed consent Pregnant or nursing women, or children under age 18
* Active infections such as herpes simplex virus (HSV) Acute, untreated medical problems such as poorly-controlled diabetes, decompensated heart failure, etc.
* There are no specific contraindications to use of the laser based on skin pigmentation, sun sensitivity, history of keloids, use of specific medications, etc.
* Appropriateness for trial entry will be determined on an individual basis by the study investigators.
* Patients with ECOG Performance Status 3 will be excluded.
* Patients with ANC 1500,PLT 50, or Hgb 8.0 will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Micheletti, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- rAblative Fractional Laser for Sclerotic GVHD-Associated Joint: Range of motion limitations and joint contractures due to sclerotic GVHD across a specific joint / limb"
  CO2 Laser: Perform ablative fractional resurfacing using a 10,600nm carbon dioxide (CO2) laser targeted to thickened, sclerotic plaques causing range of motion limitation and contracture across joints.
  Ultrasound: Patients will undergo ultrasound of the planned treatment site to measure skin thickness and blood flow via Doppler ultrasound.
  Skin Biopsy: standard 4mm punch biopsy of the skin at the planned treatment site for histologic assessment of skin thickness and sclerosis.
  Photography: Photography of the affected area / intended treatment area.
Period: Overall Study
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
Started | 8
Completed | 6
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Show Improvement in Range of Motion, Flexion, and Extension
Description: Range of motion (flexion, extension, supination, pronation) of the target joint (measured in degrees, using a goniometer).
Time Frame: 5 months from time point zero / baseline
Measure: Count of Participants; unit: Participants
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
Number analyzed (Participants) | 6
Participants | 6

2. Primary Outcome: Number of Subjects With Evidence of Collagen Remodeling (Increased Dermal Echogenicity) Compared to Baseline
Description: Measurement of skin echogencity (brightness) in comparison with pre-therapy images of the same areas using high-resolution ultrasound.
Time Frame: 3 months after final laser session (5 months after time zero / baseline)
Measure: Count of Participants; unit: Participants
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
Number analyzed (Participants) | 6
Participants | 6

3. Primary Outcome: Number of Subjects Who Show Decrease in Skin Thickness and Sclerosis With Collagen Remodeling as Measured by Before and After Skin Biopsies Biopsy
Description: Trichcrome stain, collagen fiber number and thickness, Herovici stain, elastic fiber length, and dermal thickness.
Time Frame: baseline and 3 months after final laser session
Measure: Count of Participants; unit: Participants
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
Number analyzed (Participants) | 6
Participants | 6

ADVERSE EVENTS:
Time Frame: 8 months
Arm/Group | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 1/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint (N=8)
Left Brachial artery clot (Cardiac disorders) | 1 (1) — Pt complained of L arm cramping beginning 1/21 was diagnosed with brachial artery clot on 1/26. Went to OR for thrombectomy. Now doing fine, anticoagulated. Please note laser treatment #1 for this study took place on 1/22 on contralateral wrist.
Biopsy site infection (Infections and infestations) | 1 (1) — Pt experienced pain at the right forearm skin biopsy site the same day of the biopsy. Later developed scant fibrinous exudate vs minimal purulent drainage, possibly representing superficial skin infection.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | rAblative Fractional Laser for Sclerotic GVHD-Associated Joint (N=8)
Pain at Treatment site (right foot) (Nervous system disorders) | 1 (1) — Pt ( has existing lower extremity neuropathy) developed pain at laser treatment site within ~1 hour of treatment. Pain was moderate to severe but transient resolved with conservative measures Treatment discontinuation for this patient due to pain.

LIMITATIONS AND CAVEATS:
Small number of study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes